CLINICAL TRIAL: NCT03925792
Title: Lifestyle Medicine for Enhancing Psychological Wellness in Police Officers: A Pilot Randomised Controlled Trial
Brief Title: Lifestyle Medicine for Enhancing Psychological Wellness in Police Officers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Collaborators: University of Melbourne (Other); University of Western Sydney (Other)
Responsible Party: Principal Investigator, Fiona YY Ho, Assistant Professor, Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: PSY006
Record Dates: First submitted 2019-04-22; First posted 2019-04-24 (Actual); Last update posted 2020-03-11 (Actual); Status verified 2020-03

CONDITIONS: Psychological Wellbeing
Keywords: lifestyle Medicine; police; mood; psychological being; mental health; body-mind; resilience
MeSH Terms: conditions — Psychological Well-Being

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment Group (Experimental): Lifestyle Medicine Group 1
  Interventions: Behavioral: Lifestyle Medicine
- Waitlist Control Group (Experimental): Lifestyle Medicine Group 2
  Interventions: Behavioral: Lifestyle Medicine

INTERVENTIONS:
Behavioral: Lifestyle Medicine — diet, sleep, exercise and mindfulness

SUMMARY:
This study will examine the feasibility and efficacy of lifestyle medicine for the enhancement of psychological wellness in police officers. The integrative lifestyle intervention is based on the "Healthy Body Healthy Mind (HBHM)" programme developed by the University of Melbourne. It includes lifestyle psychoeducation, physical activity, nutrition and diet, relaxation/ mindfulness, and sleep. These components are weaved with psychological elements such as stress management, cognitive restructuring, motivational interviewing, and goal setting strategies that are led by clinical psychologists. While lifestyle medicine has been recognised for centuries a a mean to improve physical health, the field of lifestyle medicine in the context of mental health is still in its infancy. Nevertheless, there is increasing evidence demonstrating the efficacy of individual components of lifestyle medicine (e.g. diet, physical activities, and sleep) on mood and stress management. With a well-researched lifestyle medicine programme adopted from Australia, the research team of the Chinese University of Hong Kong has customised the intervention protocol to fit the Chinese culture, and has conducted a pilot trial to test the protocol across different communities and work populations. The investigators aim to examine the effectiveness of an integration of multiple lifestyle adjustments on psychological wellness from a holistic body-mind perspective. Acknowledging that police officers are one of hte work populations with stressful work nature, it is in a hope that lifestyle medicine would be effective to facilitate stress coping and enhance the psychological wellness of police officers in the long run.

ELIGIBILITY:
Inclusion Criteria:

1. Hong Kong residents aged ≥ 18 years;
2. Cantonese language fluency;
3. Patient Health Questionnaire (PHQ-9) score ≥ 10; and
4. Willingness to provide informed consent and comply with the trial protocol.

Exclusion Criteria:

1. Pregnancy;
2. Have suicidal ideation with PHQ-9 item 9 score ≥ 2 (referral information to professional services will be provided to those who endorsed items on suicidal ideation);
3. Using medication or psychotherapy for depression;
4. Having unsafe conditions and are not recommended for exercising or a change in diet by physicians; and
5. Have major psychiatric, medical or neurocognitive disorders that make participation infeasible or interfere with the adherence to the lifestyle intervention.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2019-06-01 (Actual); Primary Completion 2019-11-30 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Change in the Patient Health Questionnaire (PHQ-9) | Baseline, 1-week post-treatment and 12-week post treatment
  The PHQ-9, a 20-item questionnaire used for screening, diagnosing, monitoring and measuring the severity of depression, which scores each of the nine DSM-IV criteria as "0" (not at all) to "3" (nearly every day).
  PHQ-9 scores of 5, 10, 15, and 20 represent mild, moderate, moderately severe and severe depression respectively.

SECONDARY OUTCOMES:
Change in Depression Anxiety Stress Scales (DASS-21) | Baseline, 1-week post-treatment and 12-week post treatment
  DASS-21 is a 21-items scales, comprises three sub-scales which measures the negative emotional states of depression, anxiety, and stress, over the past week. The DASS is based on a dimensional rather than a categorical conception of psychological disorder, thus it has no direct implications for the allocation of patients to discrete diagnostic categories. However, recommended cutoffs for conventional severity labels (normal, moderate, severe) are given in the DASS Manual.
  Depression Anxiety Stress Normal 0-9 0-7 0-14 Mild 10-13 8-9 15-18 Moderate 14-20 10-14 19-25 Severe 21-27 15-19 26-33 Ex. Severe 28+ 20+ 34+
Change in Insomnia Severity Index (ISI) | Baseline, 1-week post-treatment and 12-week post treatment
  ISI is a 7-item scale designed to evaluate perceived insomnia severity. Ratings on the 5-point Likert scale are obtained on the perceived severity of sleep-onset, sleep-maintenance, early morning awakening problems, satisfaction with current sleep pattern, interference with daily functioning, noticeably of impairment attributed to the sleep problem, and level of distress caused by the sleep problem.
  Total score categories: 0-7 indicates no clinically significant insomnia, 8-14 refers to subthreshold insomnia,15-21 represents clinical insomnia (moderate severity), and 22-28 is clinical insomnia (severe).
Brief Resilience Scale | Baseline, 1-week post-treatment and 12-week post treatment
  The BRS, originally developed by Smith and colleagues (2008), is a 6-item questionnaire rated on a 5-point Likert scale from 1 (strongly disagree) to 5 (strongly agree). Higher scores represent higher level of psychological resilience. The Chinese version of the test validated by Lai & Yue (2014) has demonstrated good psychometric properties (Cronbach's alpha > .72) and were comparable to the original version developed by Smith and colleagues.
  Total score divided by 6 and to be categorized: 1.00-2.99 indicates low resilience; 3.00-4.30 indicates normal resilience and 4.31-5.00 indicated high resilience.
Short Form (Six-Dimension) Health Survey (SF-6D) | Baseline, 1-week post-treatment and 12-week post treatment
  The SF-6D is a preference-based single index measure of health. A six-digit number represents each SF-6D health state, each digit denotes the level of one of six SF-6D dimensions: physical functioning, role limitation, social functioning, bodily pain, mental health, and vitality. The SF-6D index, scores from 0.0 (worst health state) to 1.0 (best health state).
Health-Promoting Lifestyle Profile (HPLP II) | Baseline, 1-week post-treatment and 12-week post treatment
  The 52-item HPLPII is composed of a total scale and six subscales to measure behaviors in the theorized dimensions of health-promoting lifestyle: spiritual growth, interpersonal relations, nutrition, physical activity, health responsibility, and stress management.
  Items are scored as Never (N) = 1, Sometimes (S)= 2, Often (O) = 3, Routinely (R) = 4 A score for overall health-promoting lifestyle is obtained by calculating a mean of the individual's responses to all 52 items; six subscale scores are obtained similarly by calculating a mean of the responses to subscale items. The use of means rather than sums of scale items is recommended to retain the 1 to 4 metric of item responses and to allow meaningful comparisons of scores across subscales.
Change in Sheehan Disability Scale (SDS) | Baseline, 1-week post-treatment and 12-week post treatment
  SDS is a brief, 5-item self-report tool that assesses functional impairment in work/school, social life, and family life. Representation of scores in terms of functional impairment: 0: not at all, 1-3: mildly, 4-6: moderately, 7-9: markedly, 10: extremely.
Physical activity (Fitbit Surge Fitness Superwatch) | Baseline, 1-week post-treatment and 12-week post treatment
  The Fitbit Surge, a commercially available accelerometer-based activity tracker, is used to examine patterns of physical activity and heart rate, objectively.
Change in Credibility-Expectancy Questionnaire (CEQ) | Baseline, 1-week post-treatment
  The 6-item CEQ yielded ratings of treatment credibility, acceptability/satisfaction, and expectations for success.

CONTACTS AND LOCATIONS:
Locations (1):
- The Chinese University of Hong Kong, Hong Kong, Hong Kong